CLINICAL TRIAL: NCT07055750
Title: Association Of Knee Pain With High-Impact Workouts Among Gym Participants: A Cross-Sectional Study
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1018
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Knee Pain Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Knee Pain With High-Impact Workouts — Individuals who have been attending the gym regularly for at least 3 months having knee pain will be assessed With High-Impact Workouts

SUMMARY:
Cross Sectional study design. The study was conducted at Burhan gym and fitness center, Vibe gym center lake city and Flexfit gym lake city, Lahore.

The sample size was 119 and the Sampling technique used was non-probability convenience sampling technique.

ELIGIBILITY:
Inclusion Criteria:

* Gym participants aged 18 to 45 years.
* Both males and females
* Individuals who have been attending the gym regularly for at least 3 months.
* Participants performing selected high-impact workouts (e.g., burpees, jump squats) at least 2 times per week for the past 3 months.
* Participants who do not require assistive devices for walking or mobility.
* Willingness to provide informed written consent for study participation.

Exclusion Criteria:

* Individuals with a history of knee surgery or major trauma to the lower limb within the past 6 months.
* Participants diagnosed with chronic joint conditions such as osteoarthritis or rheumatoid arthritis.
* Individuals with neurological or balance disorders affecting gait or movement.
* Those currently undergoing physiotherapy or orthopedic treatment for knee or lower limb issues.
* Pregnant women.
* Participants who miss more than 25% of their regular workout sessions in the last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Gym participants aged 18 to 45 years. Association Of Knee Pain With High-Impact Workouts Among Gym Participants
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-28 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 6 Month
  Numeric Pain Rating Scale No Pain 3 25 28 <.001 Mild pain (1 to 3) 19 13 32 Moderate Pain (4 to 6) 14 9 23 Severe pain (7 to 10) 23 13 36 Total 59 60 119

CONTACTS AND LOCATIONS:
Locations (1):
- Gyms, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No